CLINICAL TRIAL: NCT07164989
Title: A Patient-Centered Approach to Promote Oral Health Awareness and Practices Regarding Oral Hygiene in Adolescent Orthodontic Patients: A Randomized Controlled Trial Using Motivational Interviewing
Brief Title: Motivational Interviewing to Improve Oral Hygiene in Adolescent Orthodontic Patients
Acronym: MI-Ortho
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Yu-Yin Lin, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 300014350; UAB (Other: University of Alabama at Birmingham)
Record Dates: First submitted 2025-08-19; First posted 2025-09-10 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2025-12

CONDITIONS: Gingivitis; DMFT Index; Dental Plaque Index; Oral Hygiene Education Methods; Oral Hygiene Reinforcement During Fixed Orthodontic Treatment; Motivational Interview, OHI
Keywords: Motivational Interview; Oral Hygiene; Fixed Orthodontic Treatment
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into two parallel arms: one receiving motivational interviewing-based counseling sessions, and one receiving standard oral health education during orthodontic care. The intervention will occur during routine follow-up visits.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motivational Interviewing Group (Experimental): Motivational Interviewing (MI) will be conducted as the primary behavioral intervention in the study group. MI is a collaborative, patient-centered communication technique designed to enhance a patient's intrinsic motivation to adopt healthier behaviors. It involves five core processes: engaging, focusing, evoking, planning, and reviewing. These sessions aim to help patients identify their own goals and motivations related to oral hygiene and to foster a sense of autonomy and accountability.
  In this study, MI sessions will be delivered by a single trained dental professional who has previous formal training and experience conducting MI as part of earlier research. To maintain quality and consistency, a structured MI script and checklist based on established MI protocols will be used for each session. Sessions will take place at three different time points throughout the study period.
  Interventions: Behavioral: Motivational Interviewing-Based Counseling
- Standard Oral Health Education Group (Experimental): Participants in this group will receive the conventional oral hygiene education typically provided in orthodontic clinics. This includes verbal instructions and printed educational materials on topics such as toothbrushing technique, flossing with braces, and the importance of maintaining oral hygiene during orthodontic treatment. Education will be delivered by pediatric dental staff during scheduled orthodontic appointments at the same time points as the intervention group (baseline, 1-month, and 6-month visits). No motivational interviewing techniques will be used. This approach reflects routine care and serves as the comparator for evaluating the added value of MI.
  Interventions: Behavioral: Standard Oral Health Education

INTERVENTIONS:
Behavioral: Motivational Interviewing-Based Counseling — Motivational interviewing (MI) is a structured, patient-centered counseling technique that helps individuals explore and resolve ambivalence toward behavior change. In this study, MI sessions will be delivered by trained pediatric dental professionals during routine orthodontic visits. Each session will last approximately 10-15 minutes and will be guided by a standardized MI protocol, focusing on improving oral hygiene behavior and increasing personal motivation and responsibility for oral care among adolescent participants. Sessions will be conducted at multiple time points during the course of treatment.
  Arms: Motivational Interviewing Group
Behavioral: Standard Oral Health Education — Participants in this group will receive the conventional oral hygiene education typically provided in orthodontic clinics. This includes verbal instructions and printed educational materials on topics such as toothbrushing technique, flossing with braces, and the importance of maintaining oral hygiene during orthodontic treatment. Education will be delivered by pediatric dental staff during scheduled orthodontic appointments at the same time points as the intervention group (baseline, 1-month, and 6-month visits). No motivational interviewing techniques will be used. This approach reflects routine care and serves as the comparator for evaluating the added value of MI.
  Arms: Standard Oral Health Education Group

SUMMARY:
This study is being conducted to explore how motivational interviewing (MI), A patient-centered counseling method, can help improve oral health awareness and practices in adolescents undergoing orthodontic treatment. Adolescents often struggle to maintain good oral hygiene during orthodontic care, which can lead to complications such as gum disease, tooth decay, and poor treatment outcomes.

Participants in this study will receive brief, structured conversations focused on encouraging them to set goals and take responsibility for their oral health. These interviews are designed to be non-judgmental and supportive, helping the participants explore their own motivations for keeping their teeth and gums healthy during braces treatment.

The study will take place at a pediatric dentistry clinic and will involve adolescents aged approximately 14 to 19 who are receiving orthodontic care. The goal is to assess whether this type of communication improves their oral hygiene behaviors and outcomes compared to standard oral health education. Findings from this research may help pediatric dentists and orthodontists improve how they engage adolescent patients in taking care of their oral health.

DETAILED DESCRIPTION:
This study aims to assess the effectiveness of motivational interviewing (MI) in promoting oral health behaviors and awareness among adolescent orthodontic patients in a pediatric dentistry setting. Adolescents often face unique challenges in maintaining good oral hygiene during orthodontic treatment due to age-related factors such as motivation, compliance, and shifting priorities. As a result, they are at increased risk for plaque accumulation, gingival inflammation, and white spot lesions.

Motivational interviewing is a well-established, evidence-based counseling approach that focuses on enhancing an individual's intrinsic motivation to change by exploring and resolving ambivalence. It has shown promise in areas such as smoking cessation, weight management, and medication adherence, but its application in oral health-especially among adolescents-remains underutilized.

This randomized controlled trial will enroll adolescent patients between the ages of 14 and 19 who are currently undergoing fixed orthodontic treatment. Participants will be randomly assigned to either the intervention group (receiving MI-based counseling sessions at routine orthodontic appointments) or the control group (receiving standard oral health education). The MI sessions will be brief (approximately 15-20 minutes), conducted by trained pediatric dental professionals, using a structured MI script and checklist based on established MI protocols.

The study will evaluate oral health behaviors through self-reported questionnaires and objective clinical measures, including plaque index, gingival index, and oral hygiene compliance as recorded in follow-up appointments. Secondary outcomes will include participant satisfaction, perceived autonomy in health decisions, and parental involvement in oral care.

Ethical safeguards include patient consent, parental consent, and measures to protect participant confidentiality. Given the low-risk, behavioral nature of the intervention, the study does not require a Data Monitoring Committee. All data will be monitored by the Principal Investigator and reviewed periodically by the study team to ensure fidelity and safety.

The findings from this study are expected to provide valuable insights into how motivational interviewing can be implemented effectively in clinical dental settings to improve adolescent engagement and long-term oral health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents aged 14-19 years
* Currently undergoing fixed orthodontic treatment with active appliances in the mouth
* Available for three study encounters over a 6-month period
* Able to read, understand, and communicate in English without the use of a translator
* Able to provide consent, and whose parent/guardian also agrees to provide consent

Exclusion Criteria:

* Patients with systemic diseases or conditions that may impact oral health
* Patients who are expected to complete orthodontic treatment or have appliances removed within 6 months
* Individuals requiring interpreter services for participation
* Individuals unable or unwilling to provide consent (or whose guardians cannot provide consent)
* Currently enrolled in another behavioral or oral health intervention study.
* Any condition deemed by the investigators to make the participant ineligible for safe and effective participation.

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-10-28 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Improvement in Oral Hygiene as Measured by change in Plaque Index (Silness and Löe, 1964) | Up to 6 months per participant
  Description: Change in Plaque Index score from baseline to the 6-month follow-up. The Plaque Index is scored on a 0-3 scale, where 0 = no plaque, 1 = thin plaque detectable by probe or disclosing solution, 2 = moderate visible plaque, and 3 = abundant plaque. A decrease in score indicates improved oral hygiene.
  Time Frame: Up to 6 months per participant Unit of Measure: Mean Plaque Index score (0-3 scale)
Improvement in Oral Hygiene as Measured by change in Gingival Index (Silness and Löe, 1964) | Up to 6 months per participant
  Description: Change in Gingival Index score from baseline to the 6-month follow-up. The Gingival Index is scored on a 0-3 scale, where 0 = normal gingiva, 1 = mild inflammation, 2 = moderate inflammation, and 3 = severe inflammation. A decrease in score indicates improved gingival health.
  Time Frame: Up to 6 months per participant Unit of Measure: Mean Gingival Index score (0-3 scale)
Change in Decayed, Missing, and Filled Teeth Index (DMFT) | Up to 6 months per participant
  Description:
  The DMFT Index (Decayed, Missing, and Filled Teeth) is a standardized WHO measure of lifetime dental caries experience in permanent dentition. Each participant's teeth will be examined, and the number of decayed (D), missing (M, due to caries), and filled (F) teeth will be recorded. The total DMFT score is the sum of these categories, ranging from 0 (no caries experience) to 28 (all permanent teeth affected). Lower scores represent better oral health. Changes in DMFT from baseline to the 6-month follow-up will be assessed to determine the effectiveness of motivational interviewing compared to standard oral hygiene education.

SECONDARY OUTCOMES:
Self-Reported Oral Hygiene Behavior Questionnaire Score | Up to 6 months per participant
  Participants will complete a validated self-report questionnaire assessing their frequency and quality of oral hygiene practices (e.g., tooth brushing, flossing, use of interdental aids). Responses will be collected at baseline and at study completion. Improvement in self-reported oral hygiene behavior is expected in the motivational interviewing group compared to the control group. Self-Reported Oral Hygiene Behavior Questionnaire Score. Participants will complete a validated self-report questionnaire at baseline, 1 month, and 6 months. This will assess frequency and quality of oral hygiene practices (e.g., tooth brushing, flossing, use of interdental aids). Scoring: The questionnaire uses a Likert-type scale, with responses scored from 0 (least favorable behavior) to 4 (most favorable behavior). Range: Minimum = 0, Maximum = 20 (total score, depending on items used).
  Higher scores indicate better oral hygiene behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Yu Yin Lin, DDS, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB School of Dentistry/ Department of Pediatric Dentistry, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
Because this study involves adolescent participants and collects identifiable behavioral and dental health data, individual participant data (IPD) will not be shared to protect participant confidentiality. However, aggregate results from the study will be published and shared through peer-reviewed journals and presentations.

REFERENCES:
- [Background] Rigau-Gay MM, Claver-Garrido E, Benet M, Lusilla-Palacios P, Ustrell-Torrent JM. Effectiveness of motivational interviewing to improve oral hygiene in orthodontic patients: A randomized controlled trial. J Health Psychol. 2020 Nov-Dec;25(13-14):2362-2373. doi: 10.1177/1359105318793719. Epub 2018 Sep 10. PMID 30198774
- [Background] Cascaes AM, Bielemann RM, Clark VL, Barros AJ. Effectiveness of motivational interviewing at improving oral health: a systematic review. Rev Saude Publica. 2014 Feb;48(1):142-53. doi: 10.1590/s0034-8910.2014048004616. PMID 24789647
- See also: Motivational interviewing workbook for dental professionals, provides guidance for behavior change strategies in oral health care. — https://motivationalinterviewing.org/motivate-your-dental-patients-workbook
- Available data/document: "Educational resource supporting the study's behavioral intervention strategy using motivational interviewing in dental settings.": MI_Education_Link — https://motivationalinterviewing.org/motivate-your-dental-patients-workbook — Publicly available educational resource supporting the behavioral component of the study.